CLINICAL TRIAL: NCT01926288
Title: Efficacy and Safety of Entecavir Maleate Tablets in Chinese Patients With Hepatitis B
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CTTQ805-4
Record Dates: First submitted 2013-08-13; First posted 2013-08-20 (Estimated); Last update posted 2017-12-29 (Actual); Status verified 2013-08

CONDITIONS: Chronic Hepatitis B
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — entecavir

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- HBeAg positive group (Other): Entecavir maleate tablets (1) + blank Baraclude tablets (1),once a day Empty stomach (at least 2 hours after a meal or fasting), treatment for 48 weeks, then enter the open-label trial extended to 240 weeks .
  Blank maleate entecavir tablets (1) + Baraclude tablets (1),once a day Empty stomach (at least 2 hours after a meal or fasting), treatment for 48 weeks, then enter the open-label trial extended to 240 weeks .
  Interventions: Drug: Entecavir maleate tablets; Drug: blank Baraclude tablets; Drug: Blank maleate entecavir tablets; Drug: Baraclude tablets
- HBeAg-negative group (Other): Entecavir maleate tablets (1) + blank Baraclude tablets (1),once a day Empty stomach (at least 2 hours after a meal or fasting), treatment for 48 weeks, then enter the open-label trial extended to 240 weeks .
  Blank maleate entecavir tablets (1) + Baraclude tablets (1),once a day Empty stomach (at least 2 hours after a meal or fasting), treatment for 48 weeks, then enter the open-label trial extended to 240 weeks .
  Interventions: Drug: Entecavir maleate tablets; Drug: blank Baraclude tablets; Drug: Blank maleate entecavir tablets; Drug: Baraclude tablets

INTERVENTIONS:
Drug: Entecavir maleate tablets
Drug: blank Baraclude tablets
Drug: Blank maleate entecavir tablets
Drug: Baraclude tablets

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of Entecavir maleate tablets in Chinese patients with hepatitis B

ELIGIBILITY:
Inclusion Criteria:

1. Subjects diagnosed of HBeAg positive or negative chronic hepatitis B
2. Aged 18 to 70 years old，male or female
3. Patients with previously HBsAg-positive, HBeAg-positive for 24 weeks, HBV-DNA> 105copies/ml. HBeAg-negative for 24 weeks or more, HBV-DNA> 105 copies/ml.
4. 1.3 times the upper normal limit (1.3 × ULN) ≤ alanine aminotransferase (ALT) ≤ 10 × ULN.
5. Total serum bilirubin (TBIL) ≤ 2.5 × ULN.
6. Prothrombin activity (PTA) ≥ 60% or prothrombin time prolonged than normal ≤ 3 seconds).
7. WBC ≥ 3.5 × 109 / L, PLT ≥ 70 × 109 / L, serum albumin (ALB)≥ 35 g / L.
8. Creatinine (Cr) ≤ 1.5 × ULN.
9. If patients take intermittently with interferon, nucleoside (acid) analogues, α1 thymosin before enrollment with 24 weeks, the time is no more than 12 weeks.
10. Patients signed an informed consent form and compliance was good.

Exclusion Criteria:

1. Patients were infected with other viruses as HAV, HCV, HDV, HEV, CMV, EBV, HIV etc.
2. Patients with cirrhosis or liver cancer.
3. Patients have participated in another therapeutic clinical trial in 3 months.
4. Granulocyte count <1.5 × 109 / L, hemoglobin (HB)<100g / L, sera alpha-fetoprotein(AFP)> 100μg / L, patients' B ultrasonography pointed space-occupying lesions.
5. Patients with severe heart, kidney, endocrine hematopoietic system and neuropsychiatric diseases.
6. Patients with metabolic or autoimmune diseases such as systemic lupus erythematosus.
7. Pregnant woman, lactating women or those who wre allergic for study drug.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 287 (Actual)
Dates: Start 2008-10; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Compared with baseline, decline of serum HBV-DNA in the value | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Yu Yan yan, doctor, Principal Investigator — Department of Infectious Diseases,Peking University First Hospital; Shi Guang feng, doctor, Principal Investigator — Huashan Hospital; Xie Qing, doctor, Principal Investigator — Shanghai Jiaotong University Affiliated Ruijin Hospital; Tang Hong, doctor, Principal Investigator — West China Hospital; Zhang Da zhi, doctor, Principal Investigator — The Second Affiliated Hospital of Chongqing Medical University; Mao Qing, doctor, Principal Investigator — The First Affiliated Hospital Of The Third Mililary Medical University; Ning Qin, doctor, Principal Investigator — Tongji Medical College of Hust Tongji Medical College Huazhong University of Science and Technology; Li Jun, doctor, Principal Investigator — The First Affiliated Hospital with Nanjing Medical University; Sheng Ji fang, doctor, Principal Investigator — Zhejiang University; Cheng Xin fang, doctor, Principal Investigator — Beijing You An Hospital,Capital Medical University
Locations (9):
- China (9):
  - Department of Infectious Diseases,Peking University First Hospital, Beijing, Beijing Municipality
  - Beijing You An Hospital,Capital Medical University, Beijing, Beijing Municipality
  - The First Affiliated Hospital Of The Third Mililary Medical University, Chongqing, Chongqing Municipality
  - Tongji Medical College of Hust Tongji Medical College Huazhong University of Science and Technology, Wuhan, Hubei
  - The First Affiliated Hospital Of Nanjing Medical University, Nanjing, Jiangsu
  - Shanghai Jiaotong University Affiliated Ruijin Hospital, Shanghai, Shanghai Municipality
  - The Second Affiliated Hospital Of Chongqing Medical University, Chongqing, Sichuan
  - West China Hospital Of Sichuan University, Chongqing, Sichuan
  - The First Affiliated Hospital Of Zhejiang University, Hangzhou, Zhejiang

REFERENCES:
- [Derived] Xu JH, Wang S, Zhang DZ, Yu YY, Si CW, Zeng Z, Xu ZN, Li J, Mao Q, Tang H, Sheng JF, Chen XY, Ning Q, Shi GF, Xie Q, Zhang XQ, Dai J. One hundred and ninety-two weeks treatment of entecavir maleate for Chinese chronic hepatitis B predominantly genotyped B or C. World J Clin Cases. 2022 Oct 6;10(28):10085-10096. doi: 10.12998/wjcc.v10.i28.10085. PMID 36246814
- [Derived] Xu JH, Wang S, Xu ZN, Yu YY, Si CW, Zeng Z, Li J, Mao Q, Zhang DZ, Tang H, Sheng JF, Chen XY, Ning Q, Shi GF, Xie Q, Zhang XQ, Dai J. Entecavir maleate versus entecavir in Chinese chronic hepatitis B predominantly genotype B or C: Results at week 144. J Viral Hepat. 2017 Oct;24(10):877-884. doi: 10.1111/jvh.12710. Epub 2017 Aug 11. PMID 28345157
- [Derived] Li N, Xu JH, Yu M, Wang S, Si CW, Yu YY. Relationship between virological response and FIB-4 index in chronic hepatitis B patients with entecavir therapy. World J Gastroenterol. 2015 Nov 21;21(43):12421-9. doi: 10.3748/wjg.v21.i43.12421. PMID 26604649